CLINICAL TRIAL: NCT03949049
Title: Efficacy of Citicoline as Neuroprotector in Neonates Exposed to Hypoxia: A Randomized Controlled Trial
Brief Title: Citicoline as Neuroprotector in Neonates Exposed to Hypoxia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass Prof Tanta University, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: neonates tanta
Record Dates: First submitted 2019-05-11; First posted 2019-05-14 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Neonatal Hypoxia
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citacoline (Experimental): Citacoline as neuroprotector
  Interventions: Drug: Citicoline
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Citicoline — Citacoline as neuroprotector
  Other Names: citacoline
  Arms: Citacoline
Other: Placebo — placebo group
  Arms: Placebo

SUMMARY:
Citicoline as neuroprotector in neonates exposed to hypoxia: A randomized controlled trial

DETAILED DESCRIPTION:
Efficacy of Citicoline as neuroprotector in neonates exposed to hypoxia: A randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* neonates with hypoxia.

Exclusion Criteria:

* hypoxic ischemic encephalopathy

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
number of seizures | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Salamah, Lecturer, Principal Investigator — Pediatrics department - Kafr-Elsheikh university; May R Elsheikh, Lecturer, Study Chair — Pediatrics department - Tanta university
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salamah A, El Amrousy D, Elsheikh M, Mehrez M. Citicoline in hypoxic ischemic encephalopathy in neonates: a randomized controlled trial. Ital J Pediatr. 2023 May 12;49(1):55. doi: 10.1186/s13052-023-01452-5. PMID 37173784